CLINICAL TRIAL: NCT02307565
Title: Blood Pressure, Cerebral Blood Flow and Cognition in SCI
Brief Title: Blood Pressure, Cerebral Blood Flow and Cognition in Spinal Cord Injury
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Jill M. Wecht, Ed.D., Research Health Scientist, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WEC-13-066
Record Dates: First submitted 2014-03-21; First posted 2014-12-04 (Estimated); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injury
Keywords: Midodrine; Blood pressure; Orthostatic hypotension; Spinal Cord Injury; Sympathetic vascular control; Cerebral blood flow velocity; Cognition function tasks; Quality of Life; MRI; fMRI
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midodrine (Experimental): Arm 1 last 30 days. Subject will either be given midodrine or placebo to take during Arm 1.
  Interventions: Drug: Midodrine; Drug: Placebo
- Placebo (Placebo Comparator): Arm 2 is followed by a 14 day washout period. Arm 2 last 30 days. Subject will be given a drug (placebo or midodrine) to take during Arm 2.
  Interventions: Drug: Midodrine; Drug: Placebo

INTERVENTIONS:
Drug: Midodrine — Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Other Names: Midodrine or Placebo
Drug: Placebo — Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Other Names: Midodrine or Placebo

SUMMARY:
Following spinal cord injury autonomic regulation of the cardiovascular system is impaired, which results in a variety of measurable abnormalities in blood pressure. Evidence of causality has been documented in the general medical literature with findings of improved cognitive function following acute increases in blood pressure using the anti-hypotensive agent Midodrine Hydrochloride (midodrine). Additionally, a recent report documented an inverse association between blood pressure and depression suggesting that low blood pressure may confer greater risk than high blood pressure. Midodrine is a drug approved by the Food and Drug Administration to treat low blood pressure in the general population. Midodrine is not approved in the United States to treat low blood pressure in persons with spinal cord injury. Therefore, its use in this study is investigational. The first objective is to characterize the relationship between blood pressure, cerebral blood flow velocity and cognitive function after a single dose of midodrine compared to placebo. Second objective is to determine the long-term safety and efficacy of midodrine administration.

DETAILED DESCRIPTION:
Acute Study:The purpose of this research study is to measure a spinal cord injured individual's blood pressure and blood flow to the brain at rest and during thinking tasks before and after a single dose of midodrine, a drug used to treat low blood pressure (10 mg). Eligible participants will complete 2 visits to the laboratory. Visit 1, the subject will be given midodrine and Visit 2, the subject will be given a placebo. The order of the drug is random.

Observational Study:The purpose of this research study is to determine how blood pressure changes throughout the day in a spinal cord injured individual. There is no drug in this study. This study will last about 1 month and the subject will visit the laboratory 2 times, at the beginning and at the end of the month. The subject will be given a blood pressure monitor and will be asked to record his/her blood pressure at least 3 times a day. The laboratory visits will involve the participant discussing his/her monthly blood pressure recordings and experience with blood pressure monitor.

30-Day Crossover Study: The purpose of this research study is to determine the safety and efficacy of midodrine administration over a 30-day period of time. Midodrine is a drug approved by the Food and Drug Administration to treat low blood pressure in the general population. Midodrine is not approved in the United States to treat low blood pressure in persons with spinal cord injury. Therefore, its use in this study is investigational. The subject's participation will involve about 10 weeks and the subject will be asked to visit the laboratory 8 times. The subject will be asked to take midodrine for the first 30 days and after the 14 day washout period, the subject will be asked to take a placebo for 30 days. The order of the drug will be random. The subject and the study investigators will not know which drug the subject is receiving first and second during the 30 day-treatment phase. For visit 1,4, 5 and 8(Initial visits-start of new drug administration and Post Visits- end of new drug administration), the subject will complete many different thinking tasks while his/her blood pressure, heart rate and cerebral blood flow is taken. The subject will also complete quality of life surveys, autonomic dysreflexia surveys, and will take home a blood pressure monitor to continue to monitor blood pressure. For visit 2, 3, 6, and 7, the subject's blood pressure, cerebral blood flow and heart rate will be measured. Subject will also complete the autonomic dysreflexia survey.

30-Day Crossover & MRI/Functional MRI (fMRI) Study: Eligible participants will in addition to completing the 30-Day Crossover study (procedure explained above), will also complete a MRI/fMRI Visit 1, 4, and 8.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injured

* Between the ages of 18-65 years old.
* Level of injury is between C1-T12
* Primarily wheelchair dependent for ambulation
* Have a spinal cord injury that is ASIA Impairment Scale (AIS) grade of A, B or C
* Injury occurred more than 1 year ago
* Low blood pressure (Systolic BP less than 110 mmHg for males, Systolic BP less than 100 mmHg for females)
* Primary language is English
* I am right handed

Exclusion Criteria:

* Currently have an illness or infection
* Severe history of AD (more than 3 symptomatic events per week, evidence of blood pressure elevations above 140/90 mmHg,significant adverse subjective symptoms reporting)
* Hypertension or diabetes
* History of Traumatic Brain Injury (TBI)
* Neurological condition other than SCI (Alzheimer's disease, dementia, stroke, multiple sclerosis, Parkinson's disease, etc.)
* History of epilepsy or other seizure disorder
* Diagnosis of a psychiatric disorder such as post-traumatic stress disorder, schizophrenia or bipolar disorder
* Within the past 6 months, abused illicit drugs
* Pre-screen mini mental status exam score of less than 24, as rated by the researcher
* Vision is impaired- more than 20/60 in worst eye (with prescription eyewear)
* Coronary heart and/or artery disease
* Major surgery in the last 30 days
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-03; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill M Wecht, Ed.D, Principal Investigator — JJPVAMC; Trevor Dyson-Hudson, MD, Principal Investigator — Kessler Foundation
Locations (2):
- United States (2):
  - Kessler Foundation Research Center, West Orange, New Jersey
  - James J Peters VAMC, The Bronx, New York

REFERENCES:
- [Derived] Bloom O, Wecht JM, Legg Ditterline BE, Wang S, Ovechkin AV, Angeli CA, Arcese AA, Harkema SJ. Prolonged Targeted Cardiovascular Epidural Stimulation Improves Immunological Molecular Profile: A Case Report in Chronic Severe Spinal Cord Injury. Front Syst Neurosci. 2020 Oct 15;14:571011. doi: 10.3389/fnsys.2020.571011. eCollection 2020. PMID 33177997
- [Derived] Wecht JM, Weir JP, Katzelnick CG, Chiaravalloti ND, Kirshblum SC, Dyson-Hudson TA, Weber E, Bauman WA. Double-blinded, placebo-controlled crossover trial to determine the effects of midodrine on blood pressure during cognitive testing in persons with SCI. Spinal Cord. 2020 Sep;58(9):959-969. doi: 10.1038/s41393-020-0448-0. Epub 2020 Mar 17. PMID 32203065

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of participants eligible for study was only 19.
Groups:
- Midodrine/Placebo: Arm 1 last 30 days. Subject will either be given midodrine or placebo to take during Arm 1.
  Midodrine: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Placebo: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
- Placebo/Midodrine: Arm 2 lasts 30 days after a 14 day washout following Arm 1. Subject will be given a drug (placebo or midodrine) to take during Arm 2.
  Midodrine: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Placebo: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
Period: Overall Study
Arm/Group | Midodrine/Placebo | Placebo/Midodrine
Started | 8 | 11
Completed | 3 | 7
Not Completed | 5 | 4
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Midodrine/Placebo: Arm 1 last 30 days. Subject will be given midodrine during arm 1 and placebo during arm 2.
  Midodrine: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Placebo: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
- Placebo/Midodrine: Arm 2 last 30 days. Subject will be given placebo during arm 1 and midodrine during arm 2.
  Midodrine: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Placebo: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
- Total: Total of all reporting groups
Arm/Group | Midodrine/Placebo | Placebo/Midodrine | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (11.0) | 42.4 (10.2) | 41.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 5 | 6 | 11
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Seated systolic blood pressure following midodrine administration compared to placebo.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Midodrine: 30 days of midodrine
- Placebo: Arm 2 lasts 30 days after a 14 day washout following Arm 1. Subject will be given a drug (placebo or midodrine) to take during Arm 2.
  Midodrine: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
  Placebo: Each arm (2) will last 30 days with a 14 day washout in between each arm. Subjects nor the investigators will know which drug (midodrine or placebo) is administered to the subject for the first arm (30 days) and the second arm (30 days). The subjects will take a pill three times a day. Each subject will return home with a blood pressure monitor and will be asked to report his/her blood pressure at least 3 times a day and complete questionnaires based on how he/she is feeling.
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 19 | 12
mmHg | 116.3 (22.7) | 98.0 (23.3)

2. Secondary Outcome: Cerebral Blood Flow
Description: Middle cerebral artery blood flow velocity following midodrine administration compared to placebo.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: cm/sec
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 19 | 12
cm/sec | 45.08 (12.87) | 43.97 (16.70)

3. Secondary Outcome: Hopkins Verbal Learning Test
Description: Memory score on the Hopkins Verbal Learning Test following midodrine administration compared to placebo. Higher score is better, range from 0 to 36.
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Midodrine: Change in memory score following 30-days administration of midodrine
- Placebo: Change in memory score following 30-days administration of placebo
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 19 | 12
score on a scale | -3.56 (4.16) | -2.27 (6.47)

4. Secondary Outcome: Number of Hypertensive Events
Description: Number of daily systolic blood pressure recordings above 140 mmHg following midodrine administration compared to placebo.
Time Frame: 30 days
Measure: Number; unit: blood pressure recordings
Units Other Than Participants: blood pressure recordings
Groups:
- Midodrine: 30-days of midodrine administration
- Placebo: 30-days of placebo administration
Arm/Group | Midodrine | Placebo
Number analyzed (Participants) | 19 | 12
Number analyzed (blood pressure recordings) | 891 | 1070
blood pressure recordings | 112 | 50

ADVERSE EVENTS:
Time Frame: 30 days
Description: Risk of SAE is not greater than expected for the population. Risk of all-cause mortality is not greater than expected for the population.
Groups:
- Midodrine: 30 days of midodrine administration
- Placebo: 30 days of placebo administration
Arm/Group | Midodrine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/19 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midodrine (N=19) | Placebo (N=19)
Hypertensive response (Vascular disorders) | 3 (3) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | NA — UTI
Constipation (Renal and urinary disorders) | 1 (1) | NA — constipated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT02307565/Prot_SAP_ICF_000.pdf